CLINICAL TRIAL: NCT04489459
Title: Comparative Clinical Study Between Colistin-Tigecycline Combined Therapy Versus Colistin-Meropenem Combined Therapy in Treatment of Blood Stream Infections With Multidrug-Resistant Klebsiella Pneumoniae
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Salma Wagih Abdalla, Principle Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D12019
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Treatment of Blood Stream Infections Due to Multidrug-Resistant Klebsiella Pneumoniae
Keywords: Colistin; Tigecycline; Meropenem
MeSH Terms: interventions — Colistin; Meropenem; Tigecycline

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colistin-tigecycline (Active Comparator): this group received Intravenous colistin 9 MIU IV infusion over 2 hours loading dose followed by maintenance dose 4.5 MIU IV infusion over 2 hours q12 h plus Intravenous Tigecycline 100 mg IV infusion over 1 hour loading dose followed by maintenance dose 50 mg IV infusion over 1 hour q12h
  Interventions: Drug: Colistin; Drug: Tigecycline
- colistin-meropenem (Active Comparator): received Intravenous colistin 9 MIU IV infusion over 2 hours loading dose followed by maintenance dose 4.5 MIU IV infusion over 2 hours q12 h plus Intravenous meropenem 2 g IV infusion over 30 minutes q8 h
  Interventions: Drug: Colistin; Drug: Meropenem

INTERVENTIONS:
Drug: Colistin — Intravenous colistin 9 MIU IV infusion over 2 hours loading dose followed by maintenance dose 4.5 MIU IV infusion over 2 hours q12 h
  Other Names: polymixin B
Drug: Meropenem — Intravenous meropenem 2 g IV infusion over 30 minutes q8 h
  Arms: colistin-meropenem
Drug: Tigecycline — Intravenous Tigecycline 100 mg IV infusion over 1 hour loading dose followed by maintenance dose 50 mg IV infusion over 1 hour q12
  Arms: colistin-tigecycline

SUMMARY:
This prospective, comparative study is evaluating the effectiveness and adverse effects of using colistin at a loading dose of 9 million international units (MIU) followed by 4.5 MIU every 12 h (q12 h) + tigecycline at a loading dose of 100 mg followed by 50 mg every 12 h (q12 h) versus colistin + meropenem 2 g q8 h in treating blood stream infections due to multidrug-resistant (MDR) Klebsiella pneumoniae. The aims of the current study are to investigate and evaluate the therapeutic activity and side effects of Colistin-Meropenem combined therapy versus Colistin-Tigecycline combined therapy in treatment of patients with Multiple Drug Resistant (MDR)-Klebsiella pneumonia bacteraemia The primary goal is comparing 14 day mortality between critically ill patients with MDR Gram-negative Klebsiella pneumoniae infection as evaluation of the therapeutic activity of colistin - tigecycline vs. colistin - meropenem combined therapies. The secondary goal is comparing the comorbidities (nephrotoxicity, hepatotoxicity, neurotoxicity, hematological changes) between critically ill patients with MDR Gram-negative Klebsiella pneumoniae infection who will be treated with colistin - tigecycline versus colistin - meropenem combined therapies.

Method: A total of 60 patients were divided into two groups (30 patients each); the first group received Intravenous colistin 9 MIU IV infusion over 2 hours loading dose followed by maintenance dose 4.5 MIU IV infusion over 2 hours q12 h plus Intravenous Tigecycline 100 mg IV infusion over 1 hour loading dose followed by maintenance dose 50 mg IV infusion over 1 hour q12 and the second group received Intravenous colistin 9 MIU IV infusion over 2 hours loading dose followed by maintenance dose 4.5 MIU IV infusion over 2 hours q12 h plus Intravenous meropenem 2 g IV infusion over 30 minutes q8 h

ELIGIBILITY:
Inclusion Criteria:

* Patients with blood stream infection caused by MDR K. pneumoniae, as defined by Infectious Diseases Society of America (IDSA), who were hospitalised in the general ICU, confirmed with carbapenem-resistant K. pneumoniae-positive culture results from blood sample within the previous 5 days

Exclusion Criteria:

* All patients without a MDR carbapenem-resistant K. pneumoniae-positive culture isolated from the blood. In addition, the following patients are excluded: patients with a Glasgow Coma Scale (GCS) score of <9 in non-ventilated patients or <6 in ventilated patients; patients with end-stage metastatic malignant cancer; and all terminal patients with Acute Physiology and Chronic Health Evaluation (APACHE) II or Sequential Organ Failure Assessment (SOFA) scores of >34 or >15, respectively, and risk of mortality >85% or >80% on the first day of colistin administration, respectively [27,28]. Moreover, patients who received i.v. colistin combination therapies for <72 h are excluded from further analysis

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-21 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Comparing 14 day mortality between critically ill patients with MDR Gram-negative Klebsiella pneumoniae infection as evaluation of the therapeutic activity of colistin - tigecycline vs. colistin - meropenem combined therapies. | 7-14 days

SECONDARY OUTCOMES:
Comparing comorbidities:nephrotoxicity,hepatotoxicity,neurotoxicity,hematological changes between critically ill patients with MDR Gram-negative Klebsiella pneumoniae infection treated with colistin-tigecycline vs colistin-meropenem | 7-14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Qasr El Ainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Daikos GL, Petrikkos P, Psichogiou M, Kosmidis C, Vryonis E, Skoutelis A, Georgousi K, Tzouvelekis LS, Tassios PT, Bamia C, Petrikkos G. Prospective observational study of the impact of VIM-1 metallo-beta-lactamase on the outcome of patients with Klebsiella pneumoniae bloodstream infections. Antimicrob Agents Chemother. 2009 May;53(5):1868-73. doi: 10.1128/AAC.00782-08. Epub 2009 Feb 17. PMID 19223638
- [Background] Maltezou HC, Giakkoupi P, Maragos A, Bolikas M, Raftopoulos V, Papahatzaki H, Vrouhos G, Liakou V, Vatopoulos AC. Outbreak of infections due to KPC-2-producing Klebsiella pneumoniae in a hospital in Crete (Greece). J Infect. 2009 Mar;58(3):213-9. doi: 10.1016/j.jinf.2009.01.010. Epub 2009 Feb 26. PMID 19246099